CLINICAL TRIAL: NCT03366766
Title: Nivolumab Plus Cisplatin/Pemetrexed or Cisplatin/Gemcitabine as Induction in Resectable Non-Small Cell Lung Cancer
Brief Title: Nivolumab, Cisplatin, and Pemetrexed Disodium or Gemcitabine Hydrochloride in Treating Patients With Stage I-IIIA Non-small Cell Lung Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17P.556
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Non-Squamous Non-Small Cell Lung Carcinoma; Stage I Non-Small Cell Lung Cancer; Stage IA Non-Small Cell Lung Carcinoma; Stage IB Non-Small Cell Lung Carcinoma; Stage II Non-Small Cell Lung Cancer; Stage IIA Non-Small Cell Lung Carcinoma; Stage IIB Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (nivolumab, cisplatin, pemetrexed disodium) (Experimental): Patients with non-squamous lung cancer receive nivolumab IV over 30 minutes, cisplatin IV over 60-120 minutes, and pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 3 weeks for up to 9 weeks in the absence of disease progression or unacceptable toxicity
  Interventions: Biological: Nivolumab; Drug: Cisplatin; Drug: Pemetrexed Disodium
- Cohort I (nivolumab, cisplatin, gemcitabine hydrochloride) (Experimental): Patients with squamous lung cancer receive nivolumab IV over 30 minutes on day 1, cisplatin IV over 60-120 minutes on day 1, and gemcitabine hydrochloride IV over 1 hour on days 1 and 8. Courses repeat every 3 weeks for up to 9 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; NIVO; Opdivo; ONO-4538
Drug: Cisplatin — Given IV
  Other Names: (SP-4-2)-Diamminedichloroplatinum; Abiplatin; Blastolem; Briplatin; (CDDP) Cis-diammine-dichloroplatinum; Cis-dichloroammine Platinum (II); Metaplatin; Plastistil; Platinol; Platinex; Platinol-AQ VHA Plus; Peyrone's Salt
  Arms: Cohort I (nivolumab, cisplatin, pemetrexed disodium)
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
  Arms: Cohort I (nivolumab, cisplatin, pemetrexed disodium)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: Hydrochloride; Difluorodeoxycytidine Hydrochloride; Gemzar
  Arms: Cohort I (nivolumab, cisplatin, gemcitabine hydrochloride)

SUMMARY:
This phase II trial studies how well Nivolumab, Cisplatin, and Pemetrexed Disodium or Gemcitabine Hydrochloride in treating patients with stage I-IIIA non-small cell lung cancer that can be removed by surgery. Monoclonal antibodies, such as Nivolumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as Cisplatin and Pemetrexed Disodium or Gemcitabine Hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving Nivolumab, Cisplatin, and Pemetrexed Disodium or Gemcitabine Hydrochloride may work better in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate major pathologic response (mpCR) in patients with newly diagnosed and untreated non-small cell lung cancer (NSCLC) stage I-IIIA treated with three courses of induction nivolumab added to either cisplatin/pemetrexed or cisplatin/gemcitabine prior to surgery.

SECONDARY OBJECTIVES:

I. Safety. II. Complete pathologic response at all sites of disease. III. Major pathologic response rate at primary site. IV. Clinical complete response rate. V. 1 year progression free survival (PFS). VI. Overall survival.

TERTIARY OBJECTIVES:

I. To explore whether PDL1 expression is associated with treatment response. II. To explore whether there is a net change in the Th1/Th2 ratio (IFN-gamma, IL-4, IL10, etc.) or cell subset frequencies (M2 monocytes, myeloid-derived suppressor cells, etc.) within a patient's peripheral blood either at baseline or in response to treatment is associated with treatment response.

III. To explore whether exosomes or other immune related serum biomarkers change after combination therapy.

IV. To explore the predictive value of serial cell free deoxyribonucleic acid (DNA) levels and response.

V. PD-L1 assessment in tumor.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed non small cell lung cancer (NSCLC), not previously treated, with a plan to undergo surgery
* Stage I-IIIA (stage I tumors must be >= 4 cm) per AJCC 8th edition
* Tumor sample must be available for PD-L1 testing; archival tissue within 3 months of study enrollment will be used; if archival tissue is unavailable, a fresh biopsy will be taken
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* While blood cells 2000/ul or more
* Absolute neutrophil count 1500/ul or more
* Platelets 100,000/ul or more
* Hemoglobin 9 g/dl or more; (transfusion permitted)
* Bilirubin less than or equal to 1.5 x the upper limit of normal (except subjects with Gilbert syndrome, who can have total bilirubin < 3 mg/dl)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x the upper limit of normal
* Glomerular filtration rate (GFR) greater than or equal to 40 ml/min using the Cockcroft-Gault formula or serum creatinine less than or equal to 1.5 x (ULN) upper limit of normal
* Women of reproductive potential should have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 21 days of the study enrollment
* Women of reproductive potential must use highly effective contraception methods to avoid pregnancy for 23 weeks after the last dose of study drugs; "women of reproductive potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level more than 40 mIU/mL
* Men of reproductive potential who are sexually active with women of reproductive potential must use any contraceptive method with a failure rate of less than 1% per year; men who are receiving the study medications will be instructed to adhere to contraception for 31 weeks after the last dose of study drugs; men who are azoospermic do not require contraception
* All subjects must be able to comprehend and sign a written informed consent document

Exclusion Criteria:

* Patients who have participated in a study with an investigational agent or device within 2 weeks of enrollment
* Any prior radiotherapy to the lung
* Any prior treatment for NSCLC
* Epidermal growth factor receptor (EGFR) or alkaline phosphatase (ALK) activating alteration
* Any prior therapy with anti-PD-1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Any history of a sever hypersensitivity reaction to any monoclonal antibody
* Any history of allergy to the study drug components
* Any concurrent malignancies- exceptions include- basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or in situ cervical cancer that has undergone potentially curative therapy; patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 3 years post-diagnosis
* Participants with an active autoimmune disease or any other condition requiring systemic treatment with either corticosteroids within 14 days (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 30 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.• Patients with evidence of interstitial lung disease or active, non-infectious pneumonitis. Patients with a history of interstitial lung disease or non-infectious pneumonitis requiring treatment with steroids are also excluded.
* Patients with a known human immunodeficiency virus infection (HIV 1/2 antibodies) or acquired immunodeficiency syndrome (HIV/AIDS), active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Patients who have received a live vaccine within 30 days prior initiation of the systemic regimen
* Patients must not be receiving any other investigational agents
* Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial
* Women must not be pregnant (as above) or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Major pathologic response (mpCR) defined as < 10% viable tumor | Up to 63 days
  A minimax Simon two-stage design will be used. The mpCR rate and its associated score 95% confidence interval will be estimated using the methods

SECONDARY OUTCOMES:
Incidence of adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | Up to 6 months
  Safety data will be summarized descriptively.
Progression free survival | At 1 year
  The distribution of progression-free survival will be estimated using the Kaplan-Meier method.
Overall survival | Up to 6 months
  The distribution of overall survival will be estimated using the Kaplan-Meier method.
Overall clinical response | Up to 6 months
  Will be summarized by presence of baseline measurable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Axelrod, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (2):
- United States (2):
  - Abington Hospital - Jefferson Health, Abington, Pennsylvania
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/